CLINICAL TRIAL: NCT02150876
Title: SWiss Evaluation of Bioabsorbable Polymer-coated Everolimus-eluting Coronary sTent The SWEET Registry
Brief Title: SWiss Evaluation of Bioabsorbable Polymer-coated Everolimus-eluting Coronary sTent
Status: Completed | Type: Observational
Sponsor: University of Freiburg (Other)
Responsible Party: Principal Investigator, Stéphane Cook, Prof, Professor, University of Freiburg
Other Study IDs: The SWEET registry
Record Dates: First submitted 2014-05-27; First posted 2014-05-30 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Coronary Artery Disease
Keywords: DES; SDF; MACE; SYNERGY
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Bioresorbable polymer drug eluting stents (DES) are an indisputable improvement over first-generation DES with promising results on long-term adverse events. But the thicker polymer and/or strut may hinder its deliverability. Complex procedures challenge stent deliverability and stent delivery failure impacts clinical prognosis.

This registry aimed to assess the immediate performance of the third-generation Synergy everolimus-eluting stent (sEES) and its 12-month clinical follow-up in an all-comer population.

DETAILED DESCRIPTION:
All consecutive patients treated with the SYNERGY stent at our institutions were prospectively included in the SWEET registry. Baseline and procedural characteristics were collected at index procedure. Clinical follow-up was performed at 1 month and 1 year by clinic visit or follow-up call. The study end point was a composite of cardiac death (CD), myocardial infarction (MI) and target lesion revascularization (TLR) at 1 year.

ELIGIBILITY:
Inclusion Criteria:

1.Patient treated by everolimus-eluting SYNERGY® stent

Exclusion Criteria:

1. Patient or legal guardian won't give consent to use collected data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients treated with SYNERGY stents at Bern and Fribourg university hospitals and La Tour Hospital in Geneva until June 30, 2014 will be retrospectively included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
MACE | at 12 month follow up
  12-month device-oriented MACE (dMACE) as defined by ARC (cardiac death, MI and TLR).

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane P Cook, MD, Study Chair — University of Freiburg
Locations (1):
- University of Freiburg, Fribourg, Canton of Fribourg, Switzerland